CLINICAL TRIAL: NCT00582582
Title: Phase II Evaluation of Docetaxel Randomized With Doxercalciferol or Placebo in Patients With Advanced Prostate Cancer
Brief Title: Study of Docetaxel With Doxercalciferol or Placebo for Advanced Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of drug supply for doxercalciferol for this study
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Sanofi (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC 2001-484; CO01802
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2009-04

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Hormone Refractory; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; 1 alpha-hydroxyergocalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Docetaxel plus doxercalciferol
  Interventions: Drug: Docetaxel plus doxercalciferol
- B (Placebo Comparator): Docetaxel plus placebo
  Interventions: Drug: Docetaxel plus placebo

INTERVENTIONS:
Drug: Docetaxel plus doxercalciferol — Docetaxel 35mg/m2 IV weekly x3 every 4 weeks plus Doxercalciferol 10mcg orally every day
  Other Names: Taxotere; Hectoral; 1a,hydroxyvitamin D2; 1a-OH-D2; 1a-hydroxyerocalciferol; Vitamin D analog; prodrug of 1a,25-dihydroxyvitamin D2
  Arms: A
Drug: Docetaxel plus placebo — Docetaxel 35mg/m2 IV weekly x3 every 4 week cycle plus placebo taken orally every day
  Other Names: Taxotere
  Arms: B

SUMMARY:
The purpose of this research study is to find out the toxicities of doxercalciferol given in combination with docetaxel (Taxotere®), as well as to see how well this combination works in the treatment of prostate cancer.

DETAILED DESCRIPTION:
This is a multi-institutional, double-blinded, randomized study comparing docetaxel plus doxercalciferol versus docetaxel plus placebo in patients with metastatic hormone refractory prostate cancer. Docetaxel is given intravenously on days 1, 8 and 15 for every 28 day cycle and doxercalciferol or placebo is taken orally every day of the 28 day cycle. Please refer to the Eligibility Criteria below for key inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of the prostate.
* evidence of metastatic disease within 4 weeks of registration.
* Must meet ONE of the following:

  1. PSA >or= 10 ng/mL and at least one lesion on bone scan.
  2. Soft tissue metastases and/or visceral disease per CT scan.
* Must show progressing prostate cancer as seen by one of the following:

  1. At least one new lesion on bone scan,
  2. Increase in size or number of measurable disease lesions,
  3. At least 2 rising PSA measurements at least two weeks apart.
* Prior bilateral orchiectomy or on LHRH agonist therapy with a serum testosterone level of < 50.
* Must be off flutamide, nilutamide, or ketoconazole or herbal supplements used to treat prostate cancer at least 4 weeks prior to registration and bicalutamide at least 6 weeks prior to registration.
* No prior cytotoxic chemotherapy.
* WHO performance status of 0-2.
* Peripheral neuropathy must be < or = to grade 1.

Exclusion Criteria:

* A history of a radiographically confirmed kidney stone or pathologically confirmed calcium stone within the last 10 years.
* Patients can continue to take bisphosphonates during the study as long as the bisphosphonate was started at least 4 weeks prior to study entry and the patient continues to demonstrate a rising PSA
* No prior treatment with suramin, strontium or other therapeutic radioisotopes.
* No radiotherapy within the past 4 weeks.
* No known brain metastases.
* No chronic hypercalcemia (serum calcium >1.0 mg/dl above the upper limit of normal range), chronic gastrointestinal disease (malabsorption, surgery affecting absorption, chronic ulcerative colitis) or any condition that the investigator feels would put the patient at undue risk.
* Must not be taking digitalis, thiazide diuretics (or drugs in combination with thiazides) or calcium supplements within one week of treatment initiation.
* No active angina, known heart disease of New York Heart Association Class II-IV or a recent history (< 6 months) of myocardial infarction.
* Must not be taking steroids, anticonvulsants, fluoride, or lithium.
* Must not have urinary protein > 4gm/24 hours
* Must not have urinary calcium > or= 500 mg/24 hours
* No Coexistent second malignancy or history of prior malignancy within previous 5 years (excluding basal or squamous cell carcinoma of the skin that has been treated curatively).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate | At 12 weeks on study

SECONDARY OUTCOMES:
Safety | Duration of study participation through 30 days post last treatment dose

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States